CLINICAL TRIAL: NCT02478463
Title: A Phase 1, Multicompartmental Pharmacokinetic Study of Cabotegravir Long-acting in Healthy Adult Volunteers
Brief Title: Pharmacokinetic Study of Cabotegravir Long-acting in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201767
Record Dates: First submitted 2015-06-18; First posted 2015-06-23 (Estimated); Results first posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: Cabotegravir; Pharmacokinetic; Healthy Adult Volunteers; GSK1265744
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — cabotegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cabotegravir (Experimental): Subject will receive CAB 30 mg tablet once daily oral dose for 28 days (4 weeks) followed by a washout period of 14 to 42 days. After the washout, subject will receive a single dose of CAB LA 600 mg IM to gluteal region.
  Interventions: Drug: Cabotegravir tablet 30 mg once daily for 28 days.; Drug: Cabotegravir injection 3 mL (200 mg/mL) IM given once on Day 1.

INTERVENTIONS:
Drug: Cabotegravir tablet 30 mg once daily for 28 days. — GSK1265744B, lactose monohydrate, microcrystalline cellulose, hypromellose, sodium starch glycolate, magnesium stearate, Aquarius film-coating, white BP18237
Drug: Cabotegravir injection 3 mL (200 mg/mL) IM given once on Day 1. — Cabotegravir will be supplied as sterile suspension for injection 200 mg/mL vial. Each vial appears as sterile white to slightly colored suspension containing 200 mg/mL of CAB for administration by intramuscular (intragluteal) injection and will be administered as 1 × 3 mL Injections (3 mL [600 mg] total) IM given once on Day 1 of injection phase

SUMMARY:
Cabotegravir (CAB) long-acting (LA) is a promising candidate for human immunodeficiency virus (HIV) pre exposure prophylaxis (PrEP) due to its potent antiretroviral activity and infrequent dosing requirements. Currently, the CAB concentrations achieved in the anatomical sites associated with sexual HIV transmission following the proposed 600 milligram (mg) intramuscular (IM) PrEP dose are unknown. These data will enhance our understanding of CAB distribution to the anatomical mucosal tissue believed to be relevant to sexual HIV-1 transmission and supplement the data to support future PrEP clinical trial development. The primary objective is to determine the PK concentrations of CAB following LA administration in plasma and in vaginal tissue (VT), cervical tissue (CT), and cervicovaginal fluid (CVF) in healthy women and in rectal tissue (RT) and rectal fluid (RF) in healthy men and women following a single 600 mg IM dose. This will be a Phase 1, open label study in healthy subjects to assess the pharmacokinetics of CAB LA in the plasma and mucosal locations associated with sexual HIV-1 transmission: VT, CT, CVF, RT and RF. The study will consist of a screening period, a 28-day oral lead-in phase at a dose of 30 mg per day followed by a 14-42 day washout period, and a single dose of CAB LA 600 mg as an IM (intragluteal) injection with compartmental pharmacokinetic (PK) sampling for up to 12 weeks. Subjects will return for safety assessments and plasma PK sampling at Week 24 and Week 36 post-injection and undergo a follow-up/withdrawal visit at Week 52 post-injection.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the medical monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. A single repeat of a procedure or lab parameter is allowed to determine eligibility.
* Body weight >= 40 kilogram (kg) and body mass index (BMI) within the range 18.5 to 35 kg /meter square (inclusive).
* Male or female
* A female subject is eligible to participate if she is pre-menopausal, has an intact uterus and cervix, AND is not pregnant (as confirmed by a negative human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies: a) Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Documented Bilateral Oophorectomy. b)Reproductive potential and agrees to follow one of the options listed below in the GlaxoSmithKline (GSK) Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) requirements from 30 days prior to the first dose of study medication and until at least five terminal half-lives OR until any continuing pharmacologic effect has ended, whichever is longer (can be up to 66 weeks on study) after the last dose of study medication and completion of the follow-up visit. Female subjects desiring pregnancy or foresee that they might wish to become pregnant within 52 weeks of receiving a CAB LA injection must be excluded. All subjects participating in the study must be counseled on safe sexual practices including the use of effective barrier methods to minimize risk of HIV transmission.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Liver Function: ALT or AST > upper limit of normal (ULN)
* Total bilirubin >ULN (isolated total bilirubin >ULN is acceptable if total bilirubin is fractionated and direct bilirubin <35%)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Corrected QT (QTc) Interval: QTc > 450 milliseconds (msec):

NOTES: The QTc is the QT interval corrected for heart rate according to Bazette's formula (QTcB), machine-read or manually over-read. QTcB will be used to determine eligibility for an individual subject. Exclusion criteria for screening electrocardiogram (ECG) (a single repeat is allowed for eligibility determination): Heart rate (<45 and >100 beats per minute (bpm) for males and <50 and >100 bpm for females; QRS duration: >120 msec; QTc interval: >450 msec for males and females

* The subject's systolic blood pressure is outside the range of 90-140 millimeter (mm) mercury (Hg), or diastolic blood pressure is outside the range of 45-90 mmHg.
* History of clinically significant cardiovascular disease including:

Evidence of previous myocardial infarction (pathologic Q waves, S-T segment changes (except early repolarization); History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease; Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block (2nd degree [type II] or higher), Wolf Parkinson White [WPW] syndrome); Sinus pauses > 3 seconds.

* Any significant arrhythmia which, in the opinion of the principal Investigator and GSK Medical Monitor, will interfere with the safety for the individual subject. Non-sustained (>=3 consecutive ventricular ectopic beats) or sustained ventricular tachycardia.
* History of ongoing or clinically relevant seizure disorder within the previous 2 years, including subjects who have required treatment for seizures within this time period. A prior history of seizure, with a seizure free period of at least 2 years, off anti-epileptics, may be considered for enrolment if the investigator believes the risk of seizure recurrence is low. All cases of prior seizure history should be discussed with the medical monitor prior to enrolment
* Use of any concurrent prohibited medications as outlined in protocol
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 gram (g) of alcohol: 12 ounces (360 milliliter [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Inability or unwillingness to comply with lifestyle and/or dietary restrictions outlined in protocol.
* High-risk behavior for HIV infection which includes, but is not limited to, one of the following risk factors within six months before entering the study (Day 1 of the oral lead-in): Unprotected vaginal or anal sex with a known HIV infected person or a casual partner, engaged in sex work for money or drugs, acquired a sexually transmitted disease, high risk partner currently or in the previous six months or intravenous drug use.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* For subjects participating in magnetic resonance imaging (MRI) imaging: Contraindication for MRI scanning (as assessed by local MRI safety questionnaire), which includes but is not limited to: a) Intracranial aneurysm clips (except Sugita) or other non-MRI compatible metallic objects; b) Intra- orbital metal fragments that have not been removed by a medical professional; c) Pacemakers or other implanted cardiac rhythm management devices and non-MRI compatible heart valves, d) Inner ear implants, e) History of claustrophobia
* Positive hepatitis B surface antigen or positive hepatitis B core antibody with negative hepatitis B surface antibody test result at screening or within 3 months prior to first dose of study treatment.
* Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment
* A positive pre-study drug/alcohol screen. A positive drug screen is permitted if due to a prescribed medication, provided that medication is not on the list of prohibited medications and approved by the investigator and medical monitor.
* A positive test for HIV antibody.
* A positive pre-study screen for sexually transmitted diseases including Neisseria gonorrhea or Chlamydia trachomatis, Trichomonas, syphilis, or an active Herpes simplex virus (HSV) genital lesion.
* Presence of a tattoo or other dermatological condition overlying the buttocks which in the opinion of the investigator may interfere with the interpretation of injection site reactions.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.

Additional Criteria for Female Subjects Only:

* Any current medical conditions that in the opinion of the investigator may compromise the conduct or analysis of the genital tract sampling (e.g., active genital tract infection or lesions).
* Inability to abstain from the use of intravaginal products (e.g. tampons, spermicides, lubricants, vaginal hygiene products, diaphragms) for 72 hours prior to the genital tract sample collection visits and for up to 72 hours after.
* Inability to abstain from any sexual activity (e.g., vaginal intercourse, masturbation, and penetration of the vagina by penises, fingers, tampons, sex toys) for 72 hours prior to the genital tract sample collection visits and for up to 72 hours after.

Additional Criteria for Male Subjects and Female Subjects who consent to rectal PK sampling:

* Any current medical conditions that in the opinion of the investigator may compromise the conduct or analysis of the rectal compartment sampling (e.g., active rectal compartment infection, lesions or disease).
* Inability to abstain from the use of intrarectal products (e.g., suppositories, lubricants) for 72 hours prior to the rectal compartment sample collection visits and for up to 72 hours after.
* Inability to abstain from any receptive anal sexual activity (e.g., anal receptive intercourse and penetration of the rectum by fingers, sex toys or other) for 72 hours prior to the rectal compartment sample collection visit and for up to 72 hours after.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (2):
- United States (2):
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 1, open label study in healthy participants to assess the pharmacokinetics of cabotegravir (CAB) long-acting (LA) in the blood plasma and anatomical tissues and secretions associated with sexual human immunodeficiency virus (HIV)-1 transmission. The study was conducted across two centers in the United States.
Pre-assignment Details: A total of 29 participants were screened, of which 10 failed screening. A total of 19 participants were enrolled in the study and received study treatment.
Groups:
- Cabotegravir Oral 30 mg Followed by Cabotegravir IM 600 mg: Participants received once daily oral dose of 30 milligram (mg) cabotegravir for 28 days during the oral lead-in phase in Period 1 followed by a single intramuscular (IM) dose of 600 mg cabotegravir in Period 2. There was a washout period of up to 42 days between the two treatment periods.
Period: Treatment Period 1 (Up to Day 29)
Arm/Group | Cabotegravir Oral 30 mg Followed by Cabotegravir IM 600 mg
Started | 19
Completed | 18
Not Completed | 1
Not completed — Physician Decision | 1
Period: Washout Period (Up to 42 Days)
Arm/Group | Cabotegravir Oral 30 mg Followed by Cabotegravir IM 600 mg
Started | 18
Completed | 17
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Treatment Period 2 (Up to 52 Weeks)
Arm/Group | Cabotegravir Oral 30 mg Followed by Cabotegravir IM 600 mg
Started | 17
Completed | 16
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cabotegravir Oral 30 mg Followed by Cabotegravir IM 600 mg
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.3 (9.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - South East Asian Heritage | 1
  Black or African American | 6
  White - White/Caucasian/European Heritage | 12

OUTCOME MEASURES:

1. Primary Outcome: Cabotegravir Concentration in Blood Plasma Following IM Administration
Description: Blood samples were collected to measure cabotegravir concentration in blood plasma following a single 600 mg IM dose at indicated time-points. Evaluable Pharmacokinetic (PK) Plasma Parameter Summary Population comprised of all participants who underwent plasma PK sampling following oral dose in treatment period 1 and IM injection in treatment period 2 and had evaluable PK parameters estimated and no major protocol deviation.
Time Frame: Day 1: Pre-dose and 4 hours; one sample on Days 3, 5, 8, Weeks 4, 8, 12, 24, 36 and 52 post-dose
Population: Evaluable PK Plasma Parameter Summary Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Groups:
- Cabotegravir IM 600 mg: All participants received single IM dose of 600 mg cabotegravir in Period 2.
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 15
Micrograms per milliliter
  Day 1: Pre-dose, n=15 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than 30% values were imputed i.e. NQ assigned zero concentration) which affected the calculation.
  Day 1: 4 hours, n=15 | 0.2864 (0.10463)
  Day 3, n=15 | 3.2748 (1.74419)
  Day 5, n=15 | 5.1071 (3.09180)
  Day 8, n=15 | 5.0433 (2.92704)
  Week 4, n=15 | 2.5583 (1.00963)
  Week 8, n=15 | 0.9683 (0.73601)
  Week 12, n=15 | 0.3925 (0.40471)
  Week 24, n=15 | 0.0550 (NA) — NA indicates that standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than 30% values were imputed i.e. NQ assigned zero concentration) which affected the calculation.
  Week 36, n=15 | 0.0213 (NA) — NA indicates that standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than 30% values were imputed i.e. NQ assigned zero concentration) which affected the calculation.
  Week 52, n=14: number analyzed (Participants) | 14
  Week 52, n=14 | 0.0089 (NA) — NA indicates that standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than 30% values were imputed i.e. NQ assigned zero concentration) which affected the calculation.

2. Primary Outcome: Cabotegravir Concentration in Vaginal Tissue Following IM Administration (Female Participants)
Description: Vaginal tissue samples were collected to measure cabotegravir concentration following a single 600 mg IM dose at indicated time-points. Evaluable Tissue-Fluid and PK Parameter Population (Oral plus IM) comprised of all participants who underwent sampling following oral dose in treatment period 1 and IM injection in treatment period 2 and have both evaluable PK and evaluable tissues-fluid parameters estimated in vaginal tissue/cervical tissue/cervicovaginal fluid/rectal tissue/rectal fluid.
Time Frame: One sample on Day 3 and Week 8 post-dose
Population: Evaluable Tissue-Fluid and PK Parameter Population (Oral plus IM). Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Micrograms per milliliter
  Day 3 | 0.5286 (0.48215)
  Week 8 | 0.1809 (0.14606)

3. Primary Outcome: Cabotegravir Concentration in Cervical Tissue Following IM Administration (Female Participants)
Description: Cervical tissue samples were collected to measure cabotegravir concentration following a single 600 mg IM dose at indicated time-points.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Micrograms per milliliter
  Day 3 | 0.8016 (0.70126)
  Day 8 | 0.9261 (0.85513)
  Week 4 | 0.4409 (0.29216)
  Week 8 | 0.1570 (0.14909)
  Week 12 | 0.0460 (NA) — NA indicates that standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than 30% values were imputed i.e. NQ assigned zero concentration) which affected the calculation.

4. Primary Outcome: Cabotegravir Concentration in Cervicovaginal Fluid Following IM Administration (Female Participants)
Description: Cervicovaginal fluid samples were collected to measure cabotegravir concentration following a single 600 mg IM dose at indicated time-points.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Micrograms per milliliter
  Day 3 | 0.6604 (0.91588)
  Day 8 | 0.6175 (0.59792)
  Week 4 | 0.3209 (0.37093)
  Week 8 | 0.0905 (0.14821)
  Week 12 | 0.0901 (0.18306)

5. Primary Outcome: Cabotegravir Concentration in Rectal Tissue Following IM Administration
Description: Rectal tissue samples were collected to measure cabotegravir concentration following a single 600 mg IM dose at indicated time-points.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 13
Micrograms per milliliter
  Day 3 | 0.2824 (0.17814)
  Day 8 | 0.5146 (0.26514)
  Week 4 | 0.2620 (0.10476)
  Week 8 | 0.1037 (0.10050)
  Week 12 | 0.0348 (NA) — NA indicates that standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than 30% values were imputed i.e. NQ assigned zero concentration) which affected the calculation.

6. Primary Outcome: Cabotegravir Concentration in Rectal Fluid Following IM Administration
Description: Rectal fluid samples were collected to measure cabotegravir concentration following a single 600 mg IM dose at indicated time-points.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 12
Micrograms per milliliter
  Day 3 | 1.3868 (1.88097)
  Day 8 | 3.2046 (2.68417)
  Week 4 | 5.2674 (7.99949)
  Week 8 | 0.3233 (0.22764)
  Week 12 | 0.7901 (1.75430)

7. Secondary Outcome: Ratio of Cabotegravir Concentration in Vaginal Tissue to Cabotegravir Concentration in Blood Plasma Following IM Administration (Female Participants)
Description: Vaginal tissue and blood samples were collected to measure cabotegravir concentration following cabotegravir IM dose at indicated time-points. Data for ratio of cabotegravir concentration in vaginal tissue to cabotegravir concentration in blood plasma is presented.
Time Frame: One sample on Day 3 and Week 8 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Ratio
  Day 3 | 0.128 (43.38)
  Week 8 | 0.199 (32.66)

8. Secondary Outcome: Ratio of Cabotegravir Concentration in Cervical Tissue to Cabotegravir Concentration in Blood Plasma Following IM Administration (Female Participants)
Description: Cervical tissue and blood samples were collected to measure cabotegravir concentration following cabotegravir IM dose at indicated time-points. Data for ratio of cabotegravir concentration in cervical tissue to cabotegravir concentration in blood plasma is presented.
Time Frame: One sample on Day 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Ratio
  Day 3 | 0.203 (36.14)
  Day 8 | 0.174 (44.85)
  Week 4 | 0.139 (99.93)
  Week 8 | 0.139 (59.16)
  Week 12 | 0.101 (45.10)

9. Secondary Outcome: Ratio of Cabotegravir Concentration in Cervicovaginal Fluid to Cabotegravir Concentration in Blood Plasma Following IM Administration (Female Participants)
Description: Cervicovaginal fluid and blood samples were collected to measure cabotegravir concentration following cabotegravir IM dose at indicated time-points. Data for ratio of cabotegravir concentration in cervicovaginal fluid to cabotegravir concentration in blood plasma is presented.
Time Frame: One sample on Day 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Ratio
  Day 3 | 0.116 (174.76)
  Day 8 | 0.124 (73.53)
  Week 4 | 0.073 (277.59)
  Week 8 | 0.057 (101.03)
  Week 12 | 0.082 (112.91)

10. Secondary Outcome: Ratio of Cabotegravir Concentration in Cervical Tissue to Cabotegravir Concentration in Cervicovaginal Fluid Following IM Administration (Female Participants)
Description: Cervical tissue and cervicovaginal fluid samples were collected to measure cabotegravir concentration following cabotegravir IM dose at indicated time-points. Data for ratio of cabotegravir concentration in cervical tissue to cabotegravir concentration in cervicovaginal fluid is presented.
Time Frame: One sample on Day 3, 8, Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Ratio
  Day 3 | 1.738 (118.75)
  Day 8 | 1.405 (81.10)
  Week 4 | 1.883 (172.44)
  Week 8 | 2.785 (110.92)
  Week 12 | 1.195 (105.01)

11. Secondary Outcome: Ratio of Cabotegravir Concentration in Vaginal Tissue to Cabotegravir Concentration in Cervicovaginal Fluid Following IM Administration (Female Participants)
Description: Vaginal tissue and cervicovaginal fluid samples were collected to measure cabotegravir concentration following cabotegravir IM dose at indicated time-points. Data for ratio of cabotegravir concentration in vaginal tissue to cabotegravir concentration in cervicovaginal fluid is presented.
Time Frame: One sample on Day 3 and Week 8 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Ratio
  Day 3 | 1.095 (233.20)
  Week 8 | 3.613 (115.25)

12. Secondary Outcome: Ratio of Cabotegravir Concentration in Rectal Tissue to Cabotegravir Concentration in Blood Plasma Following IM Administration
Description: Rectal tissue and blood samples were collected to measure cabotegravir concentration following cabotegravir IM dose at indicated time-points. Data for ratio of cabotegravir concentration in rectal tissue to cabotegravir concentration in blood plasma is presented.
Time Frame: One sample on Day 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 13
Ratio
  Day 3 | 0.078 (43.13)
  Day 8 | 0.105 (22.92)
  Week 4 | 0.104 (18.79)
  Week 8 | 0.096 (27.81)
  Week 12 | 0.091 (38.62)

13. Secondary Outcome: Ratio of Cabotegravir Concentration in Rectal Fluid to Cabotegravir Concentration in Blood Plasma Following IM Administration
Description: Rectal fluid and blood samples were collected to measure cabotegravir concentration following cabotegravir IM dose at indicated time-points. Data for ratio of cabotegravir concentration in rectal fluid to cabotegravir concentration in blood plasma is presented.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 12
Ratio
  Day 3 | 0.286 (157.60)
  Day 8 | 0.581 (140.37)
  Week 4 | 0.460 (923.37)
  Week 8 | 0.302 (140.54)
  Week 12 | 0.514 (185.97)

14. Secondary Outcome: Ratio of Cabotegravir Concentration in Rectal Tissue to Cabotegravir Concentration in Rectal Fluid Following IM Administration
Description: Rectal tissue and rectal fluid samples were collected to measure cabotegravir concentration following cabotegravir IM dose at indicated time-points. Data for ratio of cabotegravir concentration in rectal tissue to cabotegravir concentration in rectal fluid is presented.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: Evaluable Tissue-Fluid and PK Parameter Population (Oral plus IM). Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 12
Ratio
  Day 3, n=11: number analyzed (Participants) | 11
  Day 3, n=11 | 0.271 (150.25)
  Day 8, n=12 | 0.185 (140.92)
  Week 4, n=12 | 0.230 (1082.13)
  Week 8, n=12 | 0.366 (133.20)
  Week 12, n=12 | 0.093 (294.16)

15. Secondary Outcome: Maximum Observed Concentration (Cmax) of Cabotegravir in Blood Plasma Following IM Administration
Description: Blood samples were collected to measure Cmax at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Day 1: Pre-dose, 4 hours, one sample on Days 3, 5, 8, Weeks 4, 8, 12, 24, 36, and 52 post-dose
Population: Evaluable PK Plasma Parameter Summary Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 15
Micrograms per milliliter | 5.04 (62.0)

16. Secondary Outcome: Cmax of Cabotegravir in Cervical Tissue Following IM Administration (Female Participants)
Description: Cervical tissue samples were collected to measure Cmax at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Micrograms per milliliter | 0.81 (105.0)

17. Secondary Outcome: Cmax of Cabotegravir in Cervicovaginal Fluid Following IM Administration (Female Participants)
Description: Cervicovaginal fluid samples were collected to measure Cmax at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Micrograms per milliliter | 0.55 (118.3)

18. Secondary Outcome: Cmax of Cabotegravir in Rectal Tissue Following IM Administration
Description: Rectal tissue samples were collected to measure Cmax at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 13
Micrograms per milliliter | 0.50 (47.0)

19. Secondary Outcome: Cmax of Cabotegravir in Rectal Fluid Following IM Administration
Description: Rectal fluid samples were collected to measure Cmax at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 12
Micrograms per milliliter | 3.27 (171.9)

20. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to Last Quantifiable Time Point (AUC[0-last]) for Cabotegravir in Blood Plasma Following IM Administration
Description: Blood samples were collected to measure AUC(0-last) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Day 1: Pre-dose, 4 hours, One sample on Days 3, 5, 8, Weeks 4, 8, 12, 24, 36, and 52 post-dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 15
Hours*microgram per milliliter | 3992.25 (24.5)

21. Secondary Outcome: AUC(0-last) for Cabotegravir in Cervical Tissue Following IM Administration (Female Participants)
Description: Cervical tissue samples were collected to measure AUC(0-last) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Hours*microgram per milliliter | 522.73 (77.0)

22. Secondary Outcome: AUC(0-last) of Cabotegravir in Cervicovaginal Fluid Following IM Administration (Female Participants)
Description: Cervicovaginal fluid samples were collected to measure AUC(0-last) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Hours*microgram per milliliter | 324.33 (121.4)

23. Secondary Outcome: AUC(0-last) for Cabotegravir in Rectal Tissue Following IM Administration
Description: Rectal tissue samples were collected to measure AUC(0-last) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 13
Hours*microgram per milliliter | 347.73 (35.5)

24. Secondary Outcome: AUC(0-last) for Cabotegravir in Rectal Fluid Following IM Administration
Description: Rectal fluid samples were collected to measure AUC(0-last) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 12
Hours*microgram per milliliter | 1841.23 (193.8)

25. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to Infinity (AUC[0-inf]) for Cabotegravir in Blood Plasma Following IM Administration
Description: Blood samples were collected to measure AUC(0-inf) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Day 1: Pre-dose, 4 hours, one sample on Days 3, 5, 8, Weeks 4, 8, 12, 24, 36, and 52 post-dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 14
Hours*microgram per milliliter | 4172.17 (23.9)

26. Secondary Outcome: AUC(0-inf) for Cabotegravir in Cervical Tissue Following IM Administration (Female Participants)
Description: Cervical tissue samples were collected to measure AUC(0-inf) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 1
Hours*microgram per milliliter | 695.72 (NA) — NA indicates that the data is not available since geometric coefficient of variation could not be calculated for a single participant.

27. Secondary Outcome: AUC(0-inf) for Cabotegravir in Cervicovaginal Fluid Following IM Administration (Female Participants)
Description: Cervicovaginal fluid samples were collected to measure AUC(0-inf) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 4
Hours*microgram per milliliter | 399.07 (99.9)

28. Secondary Outcome: AUC(0-inf) for Cabotegravir in Rectal Tissue Following IM Administration
Description: Rectal tissue samples were collected to measure AUC(0-inf) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 3
Hours*microgram per milliliter | 291.98 (34.6)

29. Secondary Outcome: AUC(0-inf) for Cabotegravir in Rectal Fluid Following IM Administration
Description: Rectal fluid samples were collected to measure AUC(0-inf) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 2
Hours*microgram per milliliter | 850.05 (42.7)

30. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to Week (WK) 4 (AUC[0-WK4]) for Cabotegravir in Blood Plasma Following IM Administration
Description: Blood samples were collected to measure AUC(0-WK4) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Day 1: Pre-dose, 4 hours, one sample on Days 3, 5, 8 and Week 4 post-dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 15
Hours*microgram per milliliter | 2141.91 (59.2)

31. Secondary Outcome: AUC(0-WK4) for Cabotegravir in Cervical Tissue Following IM Administration (Female Participants)
Description: Cervical tissue samples were collected to measure AUC(0-WK4) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8 and Week 4 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 6
Hours*microgram per milliliter | 277.48 (103.6)

32. Secondary Outcome: AUC(0-WK4) for Cabotegravir in Cervicovaginal Fluid Following IM Administration (Female Participants)
Description: Cervicovaginal fluid samples were collected to measure AUC(0-WK4) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8 and Week 4 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Hours*microgram per milliliter | 203.32 (125.5)

33. Secondary Outcome: AUC(0-WK4) for Cabotegravir in Rectal Tissue Following IM Administration
Description: Rectal tissue samples were collected to measure AUC(0-WK4) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8 and Week 4 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 12
Hours*microgram per milliliter | 206.28 (57.2)

34. Secondary Outcome: AUC(0-WK4) for Cabotegravir in Rectal Fluid Following IM Administration
Description: Rectal fluid samples were collected to measure AUC(0-WK4) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8 and Week 4 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 12
Hours*microgram per milliliter | 1170.49 (192.1)

35. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to Week 8 (AUC[0-WK8]) for Cabotegravir in Blood Plasma Following IM Administration
Description: Blood samples were collected to measure AUC(0-WK8) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Day 1: Pre-dose, 4 hours, one sample on Days 3, 5, 8, Weeks 4 and 8 post-dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 15
Hours*microgram per milliliter | 3213.62 (40.1)

36. Secondary Outcome: AUC(0-WK8) for Cabotegravir in Cervical Tissue Following IM Administration (Female Participants)
Description: Cervical tissue samples were collected to measure AUC(0-WK8) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4 and 8 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 4
Hours*microgram per milliliter | 364.74 (85.2)

37. Secondary Outcome: AUC(0-WK8) for Cabotegravir in Cervicovaginal Fluid Following IM Administration (Female Participants)
Description: Cervicovaginal fluid samples were collected to measure AUC(0-WK8) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4 and 8 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Hours*microgram per milliliter | 281.60 (124.8)

38. Secondary Outcome: AUC(0-WK8) for Cabotegravir in Rectal Tissue Following IM Administration
Description: Rectal tissue samples were collected to measure AUC(0-WK8) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4 and 8 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Hours*microgram per milliliter | 287.35 (38.7)

39. Secondary Outcome: AUC(0-WK8) for Cabotegravir in Rectal Fluid Following IM Administration
Description: Rectal fluid samples were collected to measure AUC(0-WK8) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4 and 8 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 12
Hours*microgram per milliliter | 1575.54 (202.9)

40. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to Week 12 (AUC[0-WK12]) for Cabotegravir in Blood Plasma Following IM Administration
Description: Blood samples were collected to measure AUC(0-WK12) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Day 1: Pre-dose, 4 hours, one sample on Days 3, 5, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 14
Hours*microgram per milliliter | 3639.01 (35.6)

41. Secondary Outcome: AUC(0-WK12) for Cabotegravir in Cervical Tissue Following IM Administration (Female Participants)
Description: Cervical tissue samples were collected to measure AUC(0-WK12) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 3
Hours*microgram per milliliter | 349.98 (78.9)

42. Secondary Outcome: AUC(0-WK12) for Cabotegravir in Cervicovaginal Fluid Following IM Administration (Female Participants)
Description: Cervicovaginal fluid samples were collected to measure AUC(0-WK12) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 4
Hours*microgram per milliliter | 380.92 (107.8)

43. Secondary Outcome: AUC(0-WK12) for Cabotegravir in Rectal Tissue Following IM Administration
Description: Rectal tissue samples were collected to measure AUC(0-WK12) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 4
Hours*microgram per milliliter | 323.91 (54.8)

44. Secondary Outcome: AUC(0-WK12) for Cabotegravir in Rectal Fluid Following IM Administration
Description: Rectal fluid samples were collected to measure AUC(0-WK12) at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Hours*microgram per milliliter | 1345.13 (137.7)

45. Secondary Outcome: Apparent Terminal Phase Half-life (t1/2) of Cabotegravir in Blood Plasma Following IM Administration
Description: Blood samples were collected to measure t1/2 at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Day 1: Pre-dose, 4 hours, one sample on Days 3, 5, 8, Weeks 4, 8, 12, 24, 36, and 52 post-dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 14
Hours | 459.53 (81.4)

46. Secondary Outcome: t1/2 of Cabotegravir in Cervical Tissue Following IM Administration (Female Participants)
Description: Cervical tissue samples were collected to measure t1/2 at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 1
Hours | 363.41 (NA) — NA indicates that the data is not available since geometric coefficient of variation could not be calculated for a single participant.

47. Secondary Outcome: t1/2 of Cabotegravir in Cervicovaginal Fluid Following IM Administration (Female Participants)
Description: Cervicovaginal fluid samples were collected to measure t1/2 at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 4
Hours | 355.83 (79.4)

48. Secondary Outcome: t1/2 of Cabotegravir in Rectal Tissue Following IM Administration
Description: Rectal tissue samples were collected to measure t1/2 at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 3
Hours | 567.48 (23.3)

49. Secondary Outcome: t1/2 of Cabotegravir in Rectal Fluid Following IM Administration
Description: Rectal fluid samples were collected to measure t1/2 at indicated time-points. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 2
Hours | 306.58 (3.5)

50. Secondary Outcome: Ratio of AUC(0-last) in Cervical Tissue to AUC(0-last) in Blood Plasma for Cabotegravir Following IM Administration (Female Participants)
Description: Cervical tissue and blood samples were collected to measure AUC(0-last) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-last) in cervical tissue to AUC(0-last) in blood plasma is presented.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Ratio | 0.1215 (64.86)

51. Secondary Outcome: Ratio of AUC(0-last) in Rectal Tissue to AUC(0-last) in Blood Plasma for Cabotegravir Following IM Administration
Description: Rectal tissue and blood samples were collected to measure AUC(0-last) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-last) in rectal tissue to AUC(0-last) in blood plasma is presented.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 13
Ratio | 0.0849 (21.13)

52. Secondary Outcome: Ratio of AUC(0-inf) in Cervical Tissue to AUC(0-inf) in Blood Plasma for Cabotegravir Following IM Administration (Female Participants)
Description: Cervical tissue and blood samples were collected to measure AUC(0-inf) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-inf) in cervical tissue to AUC(0-inf) in blood plasma is presented.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 1
Ratio | 0.1943 (NA) — NA indicates that the data is not available since geometric coefficient of variation could not be calculated for a single participant.

53. Secondary Outcome: Ratio of AUC(0-inf) in Rectal Tissue to AUC(0-inf) in Blood Plasma for Cabotegravir Following IM Administration
Description: Rectal tissue and blood samples were collected to measure AUC(0-inf) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-inf) in rectal tissue to AUC(0-inf) in blood plasma is presented.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 3
Ratio | 0.0766 (42.26)

54. Secondary Outcome: Ratio of AUC(0-Wk4) in Cervical Tissue to AUC(0-Wk4) in Blood Plasma for Cabotegravir Following IM Administration (Female Participants)
Description: Cervical tissue and blood samples were collected to measure AUC(0-WK4) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-WK4) in cervical tissue to AUC(0-WK4) in blood plasma is presented.
Time Frame: One sample on Days 3, 8 and Week 4 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 6
Ratio | 0.1553 (50.33)

55. Secondary Outcome: Ratio of AUC(0-Wk 4) in Rectal Tissue to AUC(0-Wk 4) in Blood Plasma for Cabotegravir Following IM Administration
Description: Rectal tissue and blood samples were collected to measure AUC(0-WK4) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-WK4) in rectal tissue to AUC(0-WK4) in blood plasma is presented.
Time Frame: One sample on Days 3, 8 and Week 4 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 12
Ratio | 0.1000 (19.30)

56. Secondary Outcome: Ratio of AUC(0-WK8) in Cervical Tissue to AUC(0-WK8) in Blood Plasma for Cabotegravir Following IM Administration (Female Participants)
Description: Cervical tissue and blood samples were collected to measure AUC(0-WK8) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-WK8) in cervical tissue to AUC(0-WK8) in blood plasma is presented.
Time Frame: One sample on Days 3, 8, Weeks 4 and 8 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 4
Ratio | 0.1492 (52.30)

57. Secondary Outcome: Ratio of AUC(0-WK8) in Rectal Tissue to AUC(0-WK8) in Blood Plasma for Cabotegravir Following IM Administration
Description: Rectal tissue and blood samples were collected to measure AUC(0-WK8) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-WK8) in rectal tissue to AUC(0-WK8) in blood plasma is presented.
Time Frame: One sample on Days 3, 8, Weeks 4 and 8 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Ratio | 0.1062 (17.46)

58. Secondary Outcome: Ratio of AUC(0-WK12) in Cervical Tissue to AUC(0-WK12) in Blood Plasma for Cabotegravir Following IM Administration (Female Participants)
Description: Cervical tissue and blood samples were collected to measure AUC(0-WK12) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-WK12) in cervical tissue to AUC(0-WK12) in blood plasma is presented.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 3
Ratio | 0.1230 (48.22)

59. Secondary Outcome: Ratio of AUC(0-WK12) in Rectal Tissue to AUC(0-WK12) in Blood Plasma for Cabotegravir Following IM Administration
Description: Rectal tissue and blood samples were collected to measure AUC(0-WK12) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-WK12) in rectal tissue to AUC(0-WK12) in blood plasma is presented.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 4
Ratio | 0.1089 (13.50)

60. Secondary Outcome: Ratio of AUC(0-last) in Cervicovaginal Fluid to AUC(0-last) in Blood Plasma for Cabotegravir Following IM Administration-female Participants
Description: Cervicovaginal fluid and blood samples were collected to measure AUC(0-last) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-last) in cervicovaginal fluid to AUC(0-last) in blood plasma is presented.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Ratio | 0.0754 (99.37)

61. Secondary Outcome: Ratio of AUC(0-last) in Rectal Fluid to AUC(0-last) in Blood Plasma for Cabotegravir Following IM Administration
Description: Rectal fluid and blood samples were collected to measure AUC(0-last) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-last) in rectal fluid to AUC(0-last) in blood plasma is presented.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 12
Ratio | 0.4445 (204.26)

62. Secondary Outcome: Ratio of AUC(0-inf) in Cervicovaginal Fluid to AUC(0-inf) in Blood Plasma for Cabotegravir Following IM Administration (Female Participants)
Description: Cervicovaginal fluid and blood samples were collected to measure AUC(0-inf) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-inf) in cervicovaginal fluid to AUC(0-inf) in blood plasma is presented.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 4
Ratio | 0.0857 (99.10)

63. Secondary Outcome: Ratio of AUC(0-inf) in Rectal Fluid to AUC(0-inf) in Blood Plasma for Cabotegravir Following IM Administration
Description: Rectal fluid and blood samples were collected to measure AUC(0-inf) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-inf) in rectal fluid to AUC(0-inf) in blood plasma is presented.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 2
Ratio | 0.1949 (80.06)

64. Secondary Outcome: Ratio of AUC(0-WK4) in Cervicovaginal Fluid to AUC(0-WK4) in Blood Plasma for Cabotegravir Following IM Administration (Female Participants)
Description: Cervicovaginal fluid and blood samples were collected to measure AUC(0-WK4) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-WK4) in cervicovaginal fluid to AUC(0-WK4) in blood plasma is presented.
Time Frame: One sample on Days 3, 8 and Week 4 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Ratio | 0.1032 (119.71)

65. Secondary Outcome: Ratio of AUC(0-WK4) in Rectal Fluid to AUC(0-WK4) in Blood Plasma for Cabotegravir Following IM Administration
Description: Rectal fluid and blood samples were collected to measure AUC(0-WK4) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-WK4) in rectal fluid to AUC(0-WK4) in blood plasma is presented.
Time Frame: One sample on Days 3, 8 and Week 4 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 12
Ratio | 0.5452 (223.58)

66. Secondary Outcome: Ratio of AUC(0-WK8) in Cervicovaginal Fluid to AUC(0-WK8) in Blood Plasma for Cabotegravir Following IM Administration (Female Participants)
Description: Cervicovaginal fluid and blood samples were collected to measure AUC(0-WK8) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-WK8) in cervicovaginal fluid to AUC(0-WK8) in blood plasma is presented.
Time Frame: One sample on Days 3, 8, Weeks 4 and 8 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Ratio | 0.0925 (124.99)

67. Secondary Outcome: Ratio of AUC(0-WK8) in Rectal Fluid to AUC(0-WK8) in Blood Plasma for Cabotegravir Following IM Administration
Description: Rectal fluid and blood samples were collected to measure AUC(0-WK8) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-WK8) in rectal fluid to AUC(0-WK8) in blood plasma is presented.
Time Frame: One sample on Days 3, 8, Weeks 4 and 8 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 12
Ratio | 0.4845 (212.20)

68. Secondary Outcome: Ratio of AUC(0-WK12) in Cervicovaginal Fluid to AUC(0-WK12) in Blood Plasma for Cabotegravir Following IM Administration (Female Participants)
Description: Cervicovaginal fluid and blood samples were collected to measure AUC(0-WK12) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-WK12) in cervicovaginal fluid to AUC(0-WK12) in blood plasma is presented.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 4
Ratio | 0.0867 (99.56)

69. Secondary Outcome: Ratio of AUC(0-WK12) in Rectal Fluid to AUC(0-WK12) in Blood Plasma for Cabotegravir Following IM Administration
Description: Rectal fluid and blood samples were collected to measure AUC(0-WK12) following cabotegravir IM dose at indicated time-points. Data for ratio of AUC(0-WK12) in rectal fluid to AUC(0-WK12) in blood plasma is presented.
Time Frame: One sample on Days 3, 8, Weeks 4, 8 and 12 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 7
Ratio | 0.3863 (154.56)

70. Secondary Outcome: Cabotegravir Concentration in Vaginal Tissue Following Oral Administration (Female Participants)
Description: Vaginal tissue samples were collected to measure cabotegravir concentration in vaginal tissue following oral 30 mg dose at indicated time-points.
Time Frame: 24 hours post-dose on Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Groups:
- Cabotegravir Oral 30 mg: All participants received oral 30 mg dose of CAB once per day for 28 days in Period 1.
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 7
Micrograms per milliliter | 0.7477 (0.50171)

71. Secondary Outcome: Cabotegravir Concentration in Cervical Tissue Following Oral Administration (Female Participants)
Description: Cervical tissue samples were collected to measure cabotegravir concentration in cervical tissue following oral 30 mg dose at indicated time-points.
Time Frame: 24 hours post-dose on Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 7
Micrograms per milliliter | 1.1009 (0.53987)

72. Secondary Outcome: Cabotegravir Concentration in Cervicovaginal Fluid Following Oral Administration (Female Participants)
Description: Cervicovaginal fluid samples were collected to measure cabotegravir concentration in cervicovaginal fluid following oral 30 mg dose at indicated time-points.
Time Frame: 24 hours post-dose on Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 7
Micrograms per milliliter | 0.8959 (0.95662)

73. Secondary Outcome: Cabotegravir Concentration in Rectal Tissue Following Oral Administration
Description: Rectal tissue samples were collected to measure cabotegravir concentration in rectal tissue following oral 30 mg dose at indicated time-points.
Time Frame: 24 hours post-dose on Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 13
Micrograms per milliliter | 0.6104 (0.24854)

74. Secondary Outcome: Cabotegravir Concentration in Rectal Fluid Following Oral Administration
Description: Rectal fluid samples were collected to measure cabotegravir concentration in rectal fluid following oral 30 mg dose at indicated time-points.
Time Frame: 24 hours post-dose on Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 12
Micrograms per milliliter | 5.5457 (6.41639)

75. Secondary Outcome: Cabotegravir Concentration in Blood Plasma Following Oral Administration
Description: Blood samples were collected to measure cabotegravir concentration in blood plasma following oral 30 mg dose at indicated time-points.
Time Frame: 24 hours post-dose on Day 28
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 15
Micrograms per milliliter | 5.7313 (2.08899)

76. Secondary Outcome: Number of Participants With Any Non-serious Adverse Event (Non-SAE) and Serious Adverse Events (SAE) Following Oral Administration of Cabotegravir
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly or birth defect or any other situation according to medical or scientific judgment, associated with liver injury and impaired liver function was categorized as SAE. Number of participants with any non-SAE and SAE are presented.
Time Frame: Up to Day 29
Population: Safety Population comprised of all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 19
Participants
  Any Non-SAE | 10
  Any SAE | 0

77. Secondary Outcome: Number of Participants With Any Non-SAE and SAE Following IM Administration of Cabotegravir
Description: as for outcome 76
Time Frame: Up to Week 52
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 17
Participants
  Any Non-SAE | 17
  Any SAE | 2

78. Secondary Outcome: Change From Baseline in Alanine Amino Transferase (ALT), Alkaline Phosphatase (ALP) and Aspartate Amino Transferase (AST) at Indicated Time Points (Oral Dose)
Description: Blood samples were collected for the assessment of clinical chemistry parameters; ALT, ALP and AST following cabotegravir oral dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Days 14 and 29
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 18
International units per Liter
  ALT, Day 14 | 1.7 (8.98)
  ALT, Day 29 | 3.5 (10.12)
  ALP, Day 14 | -0.2 (6.44)
  ALP, Day 29 | -0.4 (3.24)
  AST, Day 14 | -0.3 (3.60)
  AST, Day 29 | 1.1 (6.14)

79. Secondary Outcome: Change From Baseline in ALT, ALP and AST at Indicated Time Points (IM Dose)
Description: Blood samples were collected for the assessment of clinical chemistry parameters; ALT, ALP and AST following cabotegravir IM dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Weeks 4, 8 and 12
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 17
International units per Liter
  ALT, Week 4, n=17 | -0.2 (4.05)
  ALT, Week 8, n=16: number analyzed (Participants) | 16
  ALT, Week 8, n=16 | -0.8 (5.33)
  ALT, Week 12, n=16: number analyzed (Participants) | 16
  ALT, Week 12, n=16 | -1.4 (3.81)
  ALP, Week 4, n=15: number analyzed (Participants) | 15
  ALP, Week 4, n=15 | 2.1 (6.39)
  ALP, Week 8, n=16: number analyzed (Participants) | 16
  ALP, Week 8, n=16 | 0.6 (8.43)
  ALP, Week 12, n=16: number analyzed (Participants) | 16
  ALP, Week 12, n=16 | 1.3 (6.57)
  AST, Week 4, n=17 | 0.1 (2.87)
  AST, Week 8, n=16: number analyzed (Participants) | 16
  AST, Week 8, n=16 | 0.1 (3.76)
  AST, Week 12, n=16: number analyzed (Participants) | 16
  AST, Week 12, n=16 | -0.1 (3.50)

80. Secondary Outcome: Change From Baseline in Creatine Kinase at Indicated Time Points (Oral Dose)
Description: Blood samples were collected for the assessment of clinical chemistry parameter; creatine kinase following cabotegravir oral dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Days 14 and 29
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 18
International units per Liter
  Day 14 | -19.9 (27.23)
  Day 29 | -8.9 (46.56)

81. Secondary Outcome: Change From Baseline in Creatine Kinase at Indicated Time Points (IM Dose)
Description: Blood samples were collected for the assessment of clinical chemistry parameter; creatine kinase following cabotegravir IM dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Weeks 8 and 12
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 16
International units per Liter
  Week 8 | 19.6 (67.42)
  Week 12 | 22.2 (92.09)

82. Secondary Outcome: Change From Baseline in Creatinine, Direct Bilirubin and Total Bilirubin at Indicated Time Points (Oral Dose)
Description: Blood samples were collected for the assessment of clinical chemistry parameters; creatinine, direct bilirubin and total bilirubin following cabotegravir oral dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Days 14 and 29
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 18
Micromoles per liter
  Creatinine, Day 14, n=18 | 0.491 (5.6500)
  Creatinine, Day 29, n=18 | -0.491 (7.0929)
  Direct bilirubin, Day 14, n=11: number analyzed (Participants) | 11
  Direct bilirubin, Day 14, n=11 | -0.311 (0.6917)
  Direct bilirubin, Day 29, n=12: number analyzed (Participants) | 12
  Direct bilirubin, Day 29, n=12 | 0.428 (0.7734)
  Total bilirubin, Day 14, n=16: number analyzed (Participants) | 16
  Total bilirubin, Day 14, n=16 | -1.282 (1.9245)
  Total bilirubin, Day 29, n=16: number analyzed (Participants) | 16
  Total bilirubin, Day 29, n=16 | 0.000 (2.7217)

83. Secondary Outcome: Change From Baseline in Creatinine, Direct Bilirubin and Total Bilirubin at Indicated Time Points (IM Dose)
Description: Blood samples were collected for the assessment of clinical chemistry parameters; creatinine, direct bilirubin and total bilirubin following cabotegravir IM dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Weeks 4, 8 and 12
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 17
Micromoles per liter
  Creatinine, Week 4, n=17 | -3.640 (8.3037)
  Creatinine, Week 8, n=16: number analyzed (Participants) | 16
  Creatinine, Week 8, n=16 | -5.525 (5.4732)
  Creatinine, Week 12, n=16: number analyzed (Participants) | 16
  Creatinine, Week 12, n=16 | -3.315 (8.4637)
  Direct bilirubin, Week 4, n=10: number analyzed (Participants) | 10
  Direct bilirubin, Week 4, n=10 | -0.171 (0.5407)
  Direct bilirubin, Week 8, n=10: number analyzed (Participants) | 10
  Direct bilirubin, Week 8, n=10 | 0.171 (1.2617)
  Direct bilirubin, Week 12, n=9: number analyzed (Participants) | 9
  Direct bilirubin, Week 12, n=9 | 0.190 (1.3368)
  Total bilirubin, Week 4, n=16: number analyzed (Participants) | 16
  Total bilirubin, Week 4, n=16 | 0.641 (3.1142)
  Total bilirubin, Week 8, n=15: number analyzed (Participants) | 15
  Total bilirubin, Week 8, n=15 | 0.114 (4.2118)
  Total bilirubin, Week 12, n=14: number analyzed (Participants) | 14
  Total bilirubin, Week 12, n=14 | 1.099 (4.5789)

84. Secondary Outcome: Change From Baseline in Albumin and Total Protein at Indicated Time Points (Oral Dose)
Description: Blood samples were collected for the assessment of clinical chemistry parameters; albumin and total protein following cabotegravir oral dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Days 14 and 29
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 18
Grams per liter
  Albumin, Day 14 | -0.6 (2.85)
  Albumin, Day 29 | -0.3 (1.53)
  Total protein, Day 14 | -1.7 (3.48)
  Total protein, Day 29 | -1.4 (2.23)

85. Secondary Outcome: Change From Baseline in Albumin and Total Protein at Indicated Time Points (IM Dose)
Description: Blood samples were collected for the assessment of clinical chemistry parameters; albumin and total protein following cabotegravir IM dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Weeks 4, 8 and 12
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 17
Grams per liter
  Albumin, Week 4, n=17 | 0.3 (2.66)
  Albumin, Week 8, n=16: number analyzed (Participants) | 16
  Albumin, Week 8, n=16 | 0.3 (2.41)
  Albumin, Week 12, n=16: number analyzed (Participants) | 16
  Albumin, Week 12, n=16 | 0.6 (2.42)
  Total protein, Week 4, n=17 | 0.2 (3.23)
  Total protein, Week 8, n=15: number analyzed (Participants) | 15
  Total protein, Week 8, n=15 | -0.1 (3.53)
  Total protein, Week 12, n=16: number analyzed (Participants) | 16
  Total protein, Week 12, n=16 | 0.5 (4.31)

86. Secondary Outcome: Change From Baseline in Calcium, Glucose, Potassium, Sodium and Urea Enzymatic Colorimetry at Indicated Time Points (Oral Dose)
Description: Blood samples were collected for the assessment of clinical chemistry parameters; calcium, glucose, potassium, sodium and urea enzymatic colorimetry (UEC) following cabotegravir oral dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Days 14 and 29
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per Liter
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 18
Millimoles per Liter
  Calcium, Day 14 | -0.027722 (0.0905221)
  Calcium, Day 29 | -0.033267 (0.0774940)
  Glucose, Day 14 | 0.391654 (0.6929202)
  Glucose, Day 29 | 0.672288 (1.0302415)
  Potassium, Day 14 | -0.05 (0.296)
  Potassium, Day 29 | -0.04 (0.241)
  Sodium, Day 14 | -0.9 (1.53)
  Sodium, Day 29 | -0.3 (2.43)
  UEC, Day 14 | -0.2975 (0.97384)
  UEC, Day 29 | -0.2578 (1.14741)

87. Secondary Outcome: Change From Baseline in Calcium, Glucose, Potassium, Sodium and UEC at Indicated Time Points (IM Dose)
Description: Blood samples were collected for the assessment of clinical chemistry parameters; calcium, glucose, potassium, sodium and UEC following cabotegravir IM dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Weeks 4, 8 and 12
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Millimoles per Liter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 17
Millimoles per Liter
  Calcium, Week 4, n=17 | -0.002935 (0.0763335)
  Calcium, Week 8, n=15: number analyzed (Participants) | 15
  Calcium, Week 8, n=15 | -0.003327 (0.0610177)
  Calcium, Week 12, n=16: number analyzed (Participants) | 16
  Calcium, Week 12, n=16 | -0.001559 (0.0666177)
  Glucose, Week 4, n=17 | -0.111020 (0.6467570)
  Glucose, Week 8, n=16: number analyzed (Participants) | 16
  Glucose, Week 8, n=16 | -0.003469 (0.8073398)
  Glucose, Week 12, n=16: number analyzed (Participants) | 16
  Glucose, Week 12, n=16 | -0.149183 (0.6402427)
  Potassium, Week 4, n=17 | -0.08 (0.260)
  Potassium, Week 8, n=16: number analyzed (Participants) | 16
  Potassium, Week 8, n=16 | -0.07 (0.236)
  Potassium, Week 12, n=16: number analyzed (Participants) | 16
  Potassium, Week 12, n=16 | 0.01 (0.379)
  Sodium, Week 4, n=17 | -0.4 (2.06)
  Sodium, Week 8, n=16: number analyzed (Participants) | 16
  Sodium, Week 8, n=16 | 0.1 (1.77)
  Sodium, Week 12, n=16: number analyzed (Participants) | 16
  Sodium, Week 12, n=16 | -0.6 (1.79)
  UEC, Week 4, n=17 | -0.5250 (1.01068)
  UEC, Week 8, n=16: number analyzed (Participants) | 16
  UEC, Week 8, n=16 | -0.6694 (1.20801)
  UEC, Week 12, n=16: number analyzed (Participants) | 16
  UEC, Week 12, n=16 | -0.3570 (1.18762)

88. Secondary Outcome: Change From Baseline in Basophil Count, Eosinophil Count, Lymphocyte Count and Monocyte Count at Indicated Time Points (Oral Dose)
Description: Blood samples were collected for the assessment of hematology parameters; basophil count, eosinophil count, lymphocyte count and monocyte count following cabotegravir oral dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Days 14 and 29
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Giga cells per Liter
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 2
Giga cells per Liter
  Basophils, Day 14, n=1: number analyzed (Participants) | 1
  Basophils, Day 14, n=1 | -0.30 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant.
  Basophils, Day 29, n=2 | -0.05 (0.212)
  Eosinophils, Day 14, n=1: number analyzed (Participants) | 1
  Eosinophils, Day 14, n=1 | 0.000 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant.
  Eosinophils, Day 29, n=2 | 0.100 (0.1414)
  Lymphocytes, Day 14, n=1: number analyzed (Participants) | 1
  Lymphocytes, Day 14, n=1 | 0.500 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant.
  Lymphocytes, Day 29, n=2 | 0.400 (0.1414)
  Monocytes, Day 14, n=1: number analyzed (Participants) | 1
  Monocytes, Day 14, n=1 | 0.000 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant.
  Monocytes, Day 29, n=2 | -0.100 (0.0000)

89. Secondary Outcome: Change From Baseline in Basophil Count, Eosinophil Count, Lymphocyte Count and Monocyte Count at Indicated Time Points (IM Dose)
Description: Blood samples were collected for the assessment of hematology parameters; basophil count, eosinophil count, lymphocyte count and monocyte count following cabotegravir IM dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Weeks 4 and 8
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Giga cells per Liter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 3
Giga cells per Liter
  Basophils, Week 4, n=3 | 0.03 (0.058)
  Basophils, Week 8, n=1: number analyzed (Participants) | 1
  Basophils, Week 8, n=1 | 0.00 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant.
  Eosinophils, Week 4, n=3 | 0.000 (0.0000)
  Eosinophils, Week 8, n=1: number analyzed (Participants) | 1
  Eosinophils, Week 8, n=1 | 0.000 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant.
  Lymphocytes, Week 4, n=3 | 0.073 (0.3607)
  Lymphocytes, Week 8, n=1: number analyzed (Participants) | 1
  Lymphocytes, Week 8, n=1 | -0.300 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant.
  Monocytes, Week 4, n=3 | -0.040 (0.2425)
  Monocytes, Week 8, n=1: number analyzed (Participants) | 1
  Monocytes, Week 8, n=1 | 0.000 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant.

90. Secondary Outcome: Change From Baseline in Total Neutrophil Count at Indicated Time Points (Oral Dose)
Description: Blood samples were collected for the assessment of hematology parameter; total neutrophils count following cabotegravir oral dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Days 14 and 29
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Giga cells per Liter
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 11
Giga cells per Liter
  Day 14, n=9: number analyzed (Participants) | 9
  Day 14, n=9 | -0.353 (0.6194)
  Day 29, n=11 | -0.565 (1.1071)

91. Secondary Outcome: Change From Baseline in Total Neutrophil Count at Indicated Time Points (IM Dose)
Description: Blood samples were collected for the assessment of hematology parameters; total neutrophil count following cabotegravir IM dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Weeks 4, 8 and 12
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Giga cells per Liter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 11
Giga cells per Liter
  Week 4, n=11 | 0.539 (0.9379)
  Week 8, n=8: number analyzed (Participants) | 8
  Week 8, n=8 | 0.010 (0.8206)
  Week 12, n=7: number analyzed (Participants) | 7
  Week 12, n=7 | -0.076 (0.7115)

92. Secondary Outcome: Change From Baseline in Platelet Count and White Blood Cell (WBC) Count at Indicated Time Points (Oral Dose)
Description: Blood samples were collected for the assessment of hematology parameters; platelet count and WBC count following cabotegravir oral dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Days 1 (post-dose), 14 and 29
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Giga cells per Liter
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 18
Giga cells per Liter
  Platelets, Day 1 (post-dose), n=1: number analyzed (Participants) | 1
  Platelets, Day 1 (post-dose), n=1 | 39.0 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant.
  Platelets, Day 14, n=17: number analyzed (Participants) | 17
  Platelets, Day 14, n=17 | -6.6 (30.83)
  Platelets, Day 29, n=18 | 8.7 (29.14)
  WBCs, Day 1, n=1: number analyzed (Participants) | 1
  WBCs, Day 1, n=1 | 2.100 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant.
  WBCs, Day 14, n=17: number analyzed (Participants) | 17
  WBCs, Day 14, n=17 | -0.056 (0.8815)
  WBCs, Day 29, n=18 | -0.263 (1.1894)

93. Secondary Outcome: Change From Baseline in Platelet Count and WBC Count at Indicated Time Points (IM Dose)
Description: Blood samples were collected for the assessment of hematology parameters; platelet count and WBC count following cabotegravir IM dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Weeks 4, 8 and 12
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Giga cells per Liter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 17
Giga cells per Liter
  Platelets, Week 4, n=17 | 11.7 (21.00)
  Platelets, Week 8, n=16: number analyzed (Participants) | 16
  Platelets, Week 8, n=16 | 12.0 (25.72)
  Platelets, Week 12, n=16: number analyzed (Participants) | 16
  Platelets, Week 12, n=16 | 7.3 (18.34)
  WBCs, Week 4, n=17 | -0.053 (1.1486)
  WBCs, Week 8, n=16: number analyzed (Participants) | 16
  WBCs, Week 8, n=16 | -0.085 (0.7777)
  WBCs, Week 12, n=16: number analyzed (Participants) | 16
  WBCs, Week 12, n=16 | -0.159 (0.9395)

94. Secondary Outcome: Change From Baseline in Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC) at Indicated Time Points (Oral Dose)
Description: Blood samples were collected for the assessment of hematology parameters; hemoglobin and MCHC following cabotegravir oral dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Days 1 (post-dose), 14 and 29
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 18
Grams per Liter
  Hemoglobin, Day 1 (post-dose), n=1: number analyzed (Participants) | 1
  Hemoglobin, Day 1 (post-dose), n=1 | -6.0 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant.
  Hemoglobin, Day 14, n=17: number analyzed (Participants) | 17
  Hemoglobin, Day 14, n=17 | -5.1 (7.60)
  Hemoglobin, Day 29, n=18 | -3.6 (6.93)
  MCHC, Day 1 (post-dose), n=1: number analyzed (Participants) | 1
  MCHC, Day 1 (post-dose), n=1 | -8.0 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant.
  MCHC, Day 14, n=17: number analyzed (Participants) | 17
  MCHC, Day 14, n=17 | -1.2 (6.93)
  MCHC, Day 29, n=18 | 1.3 (7.81)

95. Secondary Outcome: Change From Baseline in Hemoglobin and MCHC at Indicated Time Points (IM Dose)
Description: Blood samples were collected for the assessment of hematology parameters; hemoglobin and MCHC following cabotegravir IM dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Weeks 4, 8 and 12
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 17
Grams per Liter
  Hemoglobin, Week 4, n=17 | -0.8 (5.25)
  Hemoglobin, Week 8, n=16: number analyzed (Participants) | 16
  Hemoglobin, Week 8, n=16 | 0.8 (6.56)
  Hemoglobin, Week 12, n=16: number analyzed (Participants) | 16
  Hemoglobin, Week 12, n=16 | 1.4 (7.31)
  MCHC, Week 4, n=17 | 0.9 (7.39)
  MCHC, Week 8, n=16: number analyzed (Participants) | 16
  MCHC, Week 8, n=16 | -0.8 (6.33)
  MCHC, Week 12, n=16: number analyzed (Participants) | 16
  MCHC, Week 12, n=16 | 1.8 (6.84)

96. Secondary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin (MCH) at Indicated Time Points (Oral Dose)
Description: Blood samples were collected for the assessment of hematology parameter; MCH following cabotegravir oral dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Days 1 (post-dose), 14 and 29
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 18
Picograms
  Day 1 (post-dose), n=1: number analyzed (Participants) | 1
  Day 1 (post-dose), n=1 | -0.90 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant.
  Day 14, n=17: number analyzed (Participants) | 17
  Day 14, n=17 | -0.22 (0.629)
  Day 29, n=18 | -0.01 (0.567)

97. Secondary Outcome: Change From Baseline in MCH at Indicated Time Points (IM Dose)
Description: Blood samples were collected for the assessment of hematology parameter; MCH following cabotegravir IM dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Weeks 4, 8 and 12
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 17
Picograms
  Week 4, n=17 | -0.15 (0.292)
  Week 8, n=16: number analyzed (Participants) | 16
  Week 8, n=16 | -0.39 (0.584)
  Week 12, n=16: number analyzed (Participants) | 16
  Week 12, n=16 | -0.36 (0.778)

98. Secondary Outcome: Change From Baseline in Mean Corpuscle Volume (MCV) at Indicated Time Points (Oral Dose)
Description: Blood samples were collected for the assessment of hematology parameter; MCV following cabotegravir oral dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Days 1 (post-dose), 14 and 29
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 18
Femtoliters
  Day 1 (post-dose), n=1: number analyzed (Participants) | 1
  Day 1 (post-dose), n=1 | -0.20 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant.
  Day 14, n=17: number analyzed (Participants) | 17
  Day 14, n=17 | -0.40 (1.052)
  Day 29, n=18 | -0.34 (1.303)

99. Secondary Outcome: Change From Baseline in MCV at Indicated Time Points (IM Dose)
Description: Blood samples were collected for the assessment of hematology parameter; MCV following cabotegravir IM dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Weeks 4, 8 and 12
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 17
Femtoliters
  Week 4, n=17 | -0.67 (1.771)
  Week 8, n=16: number analyzed (Participants) | 16
  Week 8, n=16 | -1.03 (1.799)
  Week 12, n=16: number analyzed (Participants) | 16
  Week 12, n=16 | -1.63 (1.861)

100. Secondary Outcome: Change From Baseline in Hematocrit at Indicated Time Points (Oral Dose)
Description: Blood samples were collected for the assessment of hematology parameter; hematocrit following cabotegravir oral dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Days 1 (post-dose), 14 and 29
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 18
Proportion of red blood cells in blood
  Day 1 (post-dose), n=1: number analyzed (Participants) | 1
  Day 1 (post-dose), n=1 | -0.0060 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant.
  Day 14, n=17: number analyzed (Participants) | 17
  Day 14, n=17 | -0.0135 (0.02456)
  Day 29, n=18 | -0.0122 (0.02084)

101. Secondary Outcome: Change From Baseline in Hematocrit at Indicated Time Points (IM Dose)
Description: Blood samples were collected for the assessment of hematology parameter; hematocrit following cabotegravir IM dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Weeks 4, 8 and 12
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 17
Proportion of red blood cells in blood
  Week 4, n=17 | -0.0034 (0.01703)
  Week 8, n=16: number analyzed (Participants) | 16
  Week 8, n=16 | 0.0030 (0.02145)
  Week 12, n=16: number analyzed (Participants) | 16
  Week 12, n=16 | 0.0025 (0.02196)

102. Secondary Outcome: Change From Baseline in Red Blood Cell (RBC) Count at Indicated Time Points (Oral Dose)
Description: Blood samples were collected for the assessment of hematology parameter; RBC count following cabotegravir oral dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Days 1 (post-dose), 14 and 29
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 18
Trillion cells per liter
  Day 1 (post-dose), n=1: number analyzed (Participants) | 1
  Day 1 (post-dose), n=1 | -0.050 (NA) — NA indicates that the data is not available since standard deviation could not be calculated for a single participant.
  Day 14, n=17: number analyzed (Participants) | 17
  Day 14, n=17 | -0.126 (0.2813)
  Day 29, n=18 | -0.114 (0.2360)

103. Secondary Outcome: Change From Baseline in RBC Count at Indicated Time Points (IM Dose)
Description: Blood samples were collected for the assessment of hematology parameter; RBC count following cabotegravir IM dose at indicated time-points. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Weeks 4, 8 and 12
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 17
Trillion cells per liter
  Week 4, n=17 | -0.004 (0.1718)
  Week 8, n=16: number analyzed (Participants) | 16
  Week 8, n=16 | 0.087 (0.2129)
  Week 12, n=16: number analyzed (Participants) | 16
  Week 12, n=16 | 0.117 (0.2266)

104. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Indicated Time Points (Oral Dose)
Description: SBP and DBP were measured in a semi-supine position after approximately 10 minutes rest. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Days 14 and 29
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 18
Millimeters of mercury
  SBP, Day 14 | -1.3 (8.55)
  SBP, Day 29 | -1.0 (8.64)
  DBP, Day 14 | -0.9 (7.57)
  DBP, Day 29 | 0.5 (5.96)

105. Secondary Outcome: Change From Baseline in SBP and DBP at Indicated Time Points (IM Dose)
Description: as for outcome 104
Time Frame: Baseline (Day 1, Pre-dose), Days 3, 5, 8, Weeks 4, 8, 12, 24, 36, and 52
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 17
Millimeters of mercury
  SBP, Day 3, n=17 | 0.1 (10.15)
  SBP, Day 5, n=17 | -1.5 (10.44)
  SBP, Day 8, n=17 | 3.2 (13.18)
  SBP, Week 4, n=17 | 1.8 (12.11)
  SBP, Week 8, n=16: number analyzed (Participants) | 16
  SBP, Week 8, n=16 | 0.9 (9.23)
  SBP, Week 12, n=16: number analyzed (Participants) | 16
  SBP, Week 12, n=16 | -1.1 (11.69)
  SBP, Week 24, n=16: number analyzed (Participants) | 16
  SBP, Week 24, n=16 | 2.0 (12.88)
  SBP, Week 36, n=16: number analyzed (Participants) | 16
  SBP, Week 36, n=16 | 1.7 (11.44)
  SBP, Week 52, n=15: number analyzed (Participants) | 15
  SBP, Week 52, n=15 | 0.7 (13.08)
  DBP, Day 3, n=17 | 0.5 (4.11)
  DBP, Day 5, n=17 | -0.7 (4.69)
  DBP, Day 8, n=17 | 0.6 (5.36)
  DBP, Week 4, n=17 | -0.4 (5.20)
  DBP, Week 8, n=16: number analyzed (Participants) | 16
  DBP, Week 8, n=16 | 3.3 (5.65)
  DBP, Week 12, n=16: number analyzed (Participants) | 16
  DBP, Week 12, n=16 | 0.2 (4.46)
  DBP, Week 24, n=16: number analyzed (Participants) | 16
  DBP, Week 24, n=16 | 1.0 (4.98)
  DBP, Week 36, n=16: number analyzed (Participants) | 16
  DBP, Week 36, n=16 | 2.3 (5.47)
  DBP, Week 52, n=15: number analyzed (Participants) | 15
  DBP, Week 52, n=15 | 0.1 (9.23)

106. Secondary Outcome: Change From Baseline in Pulse Rate at Indicated Time Points (Oral Dose)
Description: Pulse rate was measured in a semi-supine position after approximately 10 minutes rest. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Days 14 and 29
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 18
Beats per minute
  Day 14 | -1.0 (5.72)
  Day 29 | 2.4 (8.23)

107. Secondary Outcome: Change From Baseline in Pulse Rate at Indicated Time Points (IM Dose)
Description: as for outcome 106
Time Frame: Baseline (Day 1, Pre-dose), Days 3, 5, 8, Weeks 4, 8, 12, 24, 36, and 52
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 17
Beats per minute
  Day 3, n=17 | -0.9 (10.51)
  Day 5, n=17 | 6.2 (7.66)
  Day 8, n=17 | 1.6 (9.06)
  Week 4, n=17 | -0.6 (7.40)
  Week 8, n=16: number analyzed (Participants) | 16
  Week 8, n=16 | -0.9 (7.85)
  Week 12, n=16: number analyzed (Participants) | 16
  Week 12, n=16 | 1.3 (11.80)
  Week 24, n=16: number analyzed (Participants) | 16
  Week 24, n=16 | 1.1 (6.87)
  Week 36, n=16: number analyzed (Participants) | 16
  Week 36, n=16 | 2.6 (11.07)
  Week 52, n=15: number analyzed (Participants) | 15
  Week 52, n=15 | 1.9 (10.59)

108. Secondary Outcome: Change From Baseline in Body Temperature at Indicated Time Points (Oral Dose)
Description: Body temperature was measured in a semi-supine position after approximately 10 minutes rest. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose (Day 1) assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose), Days 14 and 29
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 18
Degrees Celsius
  Day 14 | -0.2 (0.54)
  Day 29 | -0.1 (0.46)

109. Secondary Outcome: Change From Baseline in Body Temperature at Indicated Time Points (IM Dose)
Description: as for outcome 108
Time Frame: Baseline (Day 1, Pre-dose), Days 3, 5, 8, Weeks 4, 8, 12, 24, 36, and 52
Population: as for outcome 79
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 17
Degrees Celsius
  Day 3, n=17 | -0.0 (0.36)
  Day 5, n=17 | 0.2 (0.52)
  Day 8, n=17 | 0.0 (0.37)
  Week 4, n=17 | -0.1 (0.31)
  Week 8, n=16: number analyzed (Participants) | 16
  Week 8, n=16 | -0.0 (0.47)
  Week 12, n=16: number analyzed (Participants) | 16
  Week 12, n=16 | 0.2 (0.37)
  Week 24, n=16: number analyzed (Participants) | 16
  Week 24, n=16 | -0.0 (0.39)
  Week 36, n=16: number analyzed (Participants) | 16
  Week 36, n=16 | -0.1 (0.58)
  Week 52, n=15: number analyzed (Participants) | 15
  Week 52, n=15 | 0.1 (0.61)

110. Secondary Outcome: Number of Participants With Abnormal Urinalysis Parameters Following Oral Administration of Cabotegravir
Description: Urinalysis included assessment of pH, glucose, protein, blood and ketones by dipstick method. This analysis was not planned and data was not collected and not captured in the database.
Time Frame: Up to Day 29
Population: Safety Population. This analysis was not planned and data was not collected and not captured in the database.
Arm/Group | Cabotegravir Oral 30 mg
Number analyzed (Participants) | 0

111. Secondary Outcome: Number of Participants With Abnormal Urinalysis Parameters Following IM Administration of Cabotegravir
Description: as for outcome 110
Time Frame: Up to Week 52
Population: Safety Population. This analysis was not planned and data was not collected and not captured in the database.
Arm/Group | Cabotegravir IM 600 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Non-SAEs and SAEs were collected from the start of study treatment up to Day 29 for Period 1 (Oral dose) and up to Week 52 for Period 2 (IM dose)
Description: Non-SAE and SAEs were reported for Safety Population.
Arm/Group | Cabotegravir Oral 30 mg | Cabotegravir IM 600 mg
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/19 | 2/17
Other Adverse Events (participants affected / at risk) | 10/19 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabotegravir Oral 30 mg (N=19) | Cabotegravir IM 600 mg (N=17)
Pupils unequal (Eye disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1)
Serotonin syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabotegravir Oral 30 mg (N=19) | Cabotegravir IM 600 mg (N=17)
Injection site pain (General disorders) | 0 (0) | 15 (22)
Fatigue (General disorders) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Blood glucose increased (Investigations) | 2 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT02478463/SAP_000.pdf
  • Study Protocol (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT02478463/Prot_001.pdf